CLINICAL TRIAL: NCT04886401
Title: Retrospective Observational Study on Prediction of Response to PD-1 Immunotherapy in Patients with Non Small Cell Lung Cancer Mass Tissue Imaging HyperIONTM
Brief Title: Retrospective Observational Study on Prediction of Response to PD-1 Immunotherapy in Patients with NSCLC
Acronym: PREDICTION
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0115
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: pembrolizumab; biomarkers; multiplex imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Therapeutic antibodies that block the programmed death-ligand 1 (PD-L1)/programmed death-1 (PD-1) pathway have revolutionized immuno-oncology by inducing robust and durable responses in patients with various cancer including advanced non-small-cell lung cancer (NSCLC). However, these responses only occur in a subset of patients, even in case of PD-L1 overexpression. Elucidating the determinants of response and resistance but also of severe immune-mediated adverse events is key to improving outcomes and developing new treatment strategies. Biomarkers that predict immune checkpoint inhibitors efficacy and toxicity are urgently needed and could emerge from characterization of tumor microenvironment.

The purpose of PREDICTION project is to elucidate response and toxicity predictive immunophenotypic signatures using a new in situ multiplexed strategy with imaging mass cytometry Hyperion. Patients treated with anti-PD-1 pembrolizumab will be selected on their response and toxicity profiles. Then, tumor samples will be analysed with Hyperion technology, allowing delineation of cell subpopulations and cell-cell interactions, highlighting tumor heterogeneity and to determine correlations between response and toxicity features. The number of co-analysable markers enables global vision on the same tissue section. A better understanding of the tumor microenvironment complex system will lead to discover new predictive biomarkers potentially transferable to current practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Advanced NSCLC with PD-L1 TPS of 50% or greater
* Administration of first line pembrolizumab between January 2017 & December 2019

Exclusion Criteria:

* Auto-immune disease
* Prior exposure to immunotherapy
* First dose pembrolizumab administered after December 2019

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All-comer adults with advanced NSCLC and a PD-L1 TPS of 50% or greater, measured via IHC assays on a tumor biopsy sample, and treated with first-line pembrolizumab. Anti-PD-1 monotherapy was infused every three weeks until disease progression (according to RECIST criteria v1.1) or unacceptable toxicity, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Exclusion criteria were prior exposure to immunotherapy/chemotherapy without recent biopsy before starting pembrolizumab or unavailable/insufficient tumor tissue.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Identifying predictive biomarkers of anti-PD-1 response | 1 year
  Identifying predictive biomarkers of anti-PD-1 response by highlighting discriminant cell profiles between responder and non-responder patients

CONTACTS AND LOCATIONS:
Overall Officials: Margaux GEIER, MD, Principal Investigator — CHRU Brest
Locations (1):
- CHRU de Brest, Brest, France